CLINICAL TRIAL: NCT01353937
Title: Endogenous Progenitors Cell Therapy for Diabetic Foot Ulcers
Acronym: AMD3100
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Never Activated
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-02116
Record Dates: First submitted 2011-05-12; First posted 2011-05-16 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Diabetic Ulcer
Keywords: wound healing
MeSH Terms: interventions — plerixafor; Becaplermin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard of Care (No Intervention): All patients will be receiving the Standard of Care treatments regardless of whether or not they are receiving study drug.
- Novel Combination Therapy (Active Comparator): AMD3100 (Plerixafor) injection with Regranex Gel topical application
  Interventions: Drug: AMD3100 injection + rhPDGF-BB topical
- Becaplermin (Regranex Gel) (Active Comparator): Topical application
  Interventions: Drug: AMD3100 injection + rhPDGF-BB topical

INTERVENTIONS:
Drug: AMD3100 injection + rhPDGF-BB topical — drug therapy to be given for the first 2 week duration given on a daily basis initiated during the first visit (Day 0).
  Other Names: AMD3100 (Plerixafor); rhPDGF-BB (Becaplermin); Regranex Gel
  Arms: Becaplermin (Regranex Gel); Novel Combination Therapy

SUMMARY:
Diabetic foot ulcers, a complication of diabetes leading to 80.000 lower limb amputations annually in the US, are a significant burden to our health system, costing more than a billion dollars annually. Here, we propose a novel combination of two drugs (Mozobil® and Regranex®Gel) to mobilize a specific sub-type of stem cells (endothelial progenitor cells) from the bone marrow and traffic them toward the wound, increasing the blood supply that subsequently improves wound healing. Because we are using the human body's own resources to regenerate itself by targeting and correcting the underlying pathophysiology, we believe that this novel therapy yields great promise in the treatment of diabetic foot ulcers.

DETAILED DESCRIPTION:
Because diabetes impairs wound healing by altering fibroblast function, promotes chronic infection and diminishes blood supply to the skin, the lifetime risk of a person with diabetes developing a diabetic foot ulcer (DFU) is as high as 25%. Current strategies focus independently on the fibroblast dysfunction (growth factors such as PDGF/Regranex® Gel), on the chronic infection (debridement, antibacterial dressings) or on the blood supply (VAC®).

This project is different from the other projects because we propose to combine two drugs in a dual approach to first improve the fibroblast function using PDGF/Regranex® Gel and second to induce neovascularization in DFU by recruiting progenitor cells into the wound through a combination therapy of subcutaneous AMD3100 (Plerixafor/Mozobil®) with topical PDGF/Regranex® Gel. By contrast to novel stem cell therapies where cells are extracted, processed ex vivo and engrafted into the wound (exogenous stem cell therapy), here we propose to keep the stem cells in vivo (endogenous stem cell therapy).

Specifically, the first aim of the study will be to launch a prospective evaluator-blind pilot phase I/II safety and efficacy study to evaluate the clinical effect of AMD3100 (Plerixafor/Mozobil®) treatment with topical PDGF/Regranex® Gel compared to historical controls (standard of care and PDGF). AMD3100 (240 µg/kg SC) will be administered daily for 2 weeks. Our primary endpoint will be the measure of the percentage of change in area of the wound at 4 weeks (surrogate endpoint). In a second aim, we will measure the effect of AMD3100 treatment with PDGF using a quality-of-life index dedicated to DFU (DFS-SF).

Because we are addressing the underlying physiopathology in a dual approach, because we are avoiding the need for ex vivo processing and because both drugs are FDA approved, we believe that this novel therapy yields great promise in the treatment of DFUs.

ELIGIBILITY:
Inclusion Criteria:

1. Insulin-dependant type 2 diabetic patients
2. Age between 35 and 60 years-old
3. HbA1C between 6 and 12%
4. Full-thickness diabetic neuropathic foot ulcers
5. ≥ 2 weeks duration
6. Following standard of care débridement, ulcer size must be between 1 and 6 cm2
7. Adequate perfusion, defined as either transcutaneous oxygen measurements on the dorsum of the foot >30 mmHg or ankle brachial indexes 0.7<ABI<1.2, as well as toe pressure >30 mmHg.

Exclusion Criteria:

1. Clinical infection at the studied ulcer site (bacterial and fungal)
2. Clinically significant lower-extremity ischemia (as defined by an ankle/brachial index of <0.65)
3. Active Charcot's foot as determined by clinical and radiographic examination
4. Ulcer of a non-diabetic pathophysiology (e.g., rheumatoid, radiation-related, and vasculitis-related ulcers, and especially venous stasis ulcer)
5. Significant medical conditions that would impair wound healing will also be excluded from the study. These conditions include liver disease, aplastic anemia, scleroderma and malignancy, treatment with immunosuppressive agents or steroids, myocardial infarcts, stroke, major surgery within 6 months of the study, usage of tobacco
6. Subjects with cancerous or pre-cancerous lesions in the area to be treated
7. Body weight > 160 kg (because of Plerixafor's pharmacokinetic limitation)
8. Severe renal dysfunction (creatinine clearance < 50 ml/min)
9. Severe non-proliferative or proliferative diabetic retinopathy
10. Capillary blood glucose >350

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Rate of Wound Closure | 1 year
  The safety and efficacy of AMD3100 (Plerixafor) with rhPDGF-BB (Becaplermin) compared to two historical treatments group (Beclapermin versus standard of care (SOC) treatment) for the treatment of DFUs.[21] The central hypothesis to be tested is that a novel combination therapy will significantly increase the rate of closure of DFUs as compared to historical treatments groups, while presenting no major side effect.
Quality of Life | 4 weeks
  Test whether patients treated with the novel combination therapy will have an improvement in their quality of life, with higher scores on the DFS-SF than those of the historical control groups.

SECONDARY OUTCOMES:
Glycosylated hemoglobin (HbA1C) | 4 weeks
  long-term measure of diabetes control
capillary blood glucose (ACCUCHEK Finger Stick) | 4 weeks
  short-term measure of diabetes control
Transcutaneous oxygen tension measurements on wound and 1 cm-radius periphery (Radiometer adult sensor) | 4 weeks
  non-invasive measure of skin circulation
Ankle-brachial index (ABI, Prestige sphygmomanometer and Summit doppler probe) | 4 weeks
  measure of peripheral vascular disease
pain (Visual-Analog Scale) | 4 weeks
  measure of the subjective symptom of pain
temperature of surrounding skin in a 1 cm-radius around the DFU (TempTouch Dermal Thermometer) | 4 weeks
  to identify increased skin temperatures, intended as an early warning of inflammation, impending infection, and possible foot ulceration.
sensation (Nk Pressure-Specified Sensory Device) | 4 weeks
  Quantification of sensory nerve function in patients with symptoms of, or the potential for, neurologic damage or disease
photogrammetry (Photoshop CS3, Adobe Systems) | 4 weeks
  used to document wound appearance
glomerular filtration rate (GFR, estimated by 24 hr. urine creatinine measurement) | 4 weeks
  to estimate renal function
diabetic retinopathy (digital ophthalmologic examination) | 4 weeks
  to evaluate for development of nonproliferative and proliferative retinopathy
cEPCs by FACS analysis | 4 weeks
  to measure the extent of BM EPC mobilization into the circulation and correlate the number cEPCs to other primary and secondary endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Warren, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Helen L. & Martin S. Kimmel Wound Healing Center at the NYU Hospital for Joint Diseases, New York, New York, United States